CLINICAL TRIAL: NCT03978390
Title: Behavioral Interventions to Improve Pediatric Patients' Cooperation During the Dental Injection: a Randomized Clinical Trial
Brief Title: Improving Children's Cooperation During Dental Injection
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Change in research direction
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: Pro00091797
Record Dates: First submitted 2019-06-05; First posted 2019-06-07 (Actual); Last update posted 2020-07-27 (Actual); Status verified 2020-07

CONDITIONS: Child Behavior; Acute Pain
Keywords: Dental Injection; Behavioral Intervention; Behavioral Priming; Endowment Effect; Personality Traits
MeSH Terms: conditions — Child Behavior; Acute Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Superhero images, Reward at the beginning, (Experimental): Also, Showing superhero images for 5 minutes before starting the dental procedure. Also, providing the children with reward before begging the dental procedure and telling them that they can only keep it if they cooperate during the treatment procedure.
  Interventions: Behavioral: behavioral priming; Behavioral: endowment effect
- Superhero images, Reward at the end (Experimental): Universally-accepted positive reinforcement to increase children cooperation in dental settings
  Interventions: Behavioral: behavioral priming; Behavioral: Positive reinforcement
- No Superhero Images, Reward at the beginning (Experimental): Showing superhero images for 5 minutes before starting the dental procedure
  Interventions: Behavioral: endowment effect
- No Superhero Images, Reward at the end (Active Comparator): Showing no picture before starting the dental procedure
  Interventions: Behavioral: Positive reinforcement

INTERVENTIONS:
Behavioral: behavioral priming — Priming the children with images of superheroes in order to behave desirably during the dental injection
  Arms: Superhero images, Reward at the beginning,; Superhero images, Reward at the end
Behavioral: endowment effect — Giving the rewards to children before starting the dental treatment and telling children they can only keep it if they behave desirably during the dental procedure
  Arms: No Superhero Images, Reward at the beginning; Superhero images, Reward at the beginning,
Behavioral: Positive reinforcement — Giving rewards to the children at the end if they cooperate desirably during the treatment
  Arms: No Superhero Images, Reward at the end; Superhero images, Reward at the end

SUMMARY:
This clinical trial aims to investigate how to increase children cooperation in dental settings using ideas adopted from psychology to make an effective interdisciplinary approach. We want to test how showing images of mainstream superheroes such as Superman, Batman, etc. can prepare children, 6-12 years old, to behave desirably during the dental injection. Also, new modification will be applied to providing awards to children by telling them that they can keep the rewards they receive before starting the procedure only if they behave accordingly during the treatment. Moreover, it will be shown that if children's baseline psychological characteristic, age, gender, and family income affect their cooperation in the dental office. The results of this study help to manage children's behavior more efficiently in the clinical settings which is crucial to achieving effective treatment.

DETAILED DESCRIPTION:
Purpose:

This clinical trial aims to evaluate the impact of priming effect and endowment effect, concepts derived from psychology, on the behavior of children in mixed dentition period during the dental injection. The moderating role of the psychological traits and demographics of children will be investigated as well. The judgment on the children behaviors will be made based on a well-established instrument which categorizes the behaviors into four levels. The results will contribute to an interdisciplinary approach toward patient management and a treatment plan that let practitioners manage their time more efficiently, and also increase the chance of children's acceptable behaviors and cooperation during a dental visit and attendance in follow-up sessions.

Justification:

Patient management in pediatric dentistry is a matter of great importance as many children may not be as cooperative as adults with their dentist when undergoing dental procedures. Although there were developments in patient management in dentistry, particularly in the pediatric field, an interdisciplinary approach is still lacking to cover all aspects of behavioral management. Specifically, the findings derived from psychology and economics may have the potential to be implemented in the medical field. That being said, the concepts such as behavioral priming and endowment effect and constructs such as personality traits which have led to promising results in cognitive and behavioral management have been scarcely implemented in the medical field and dentistry.

Conditioning or contingency reinforcement is one of the universally accepted techniques in the behavioral management of children in dental clinics. The positive reinforcement is the common approach for reinforcing the desired behaviors in children. Positive reinforcement relies on promising children with positive social feedback (e.g., smile and praise) or non-social token and rewards (e.g., badges and stickers). Although positive reinforcement was reported to be successful, according to the concept of the endowment effect, other conditions of providing awards to children may be even more efficient. The endowment effect, which is a well-reported psychological phenomenon, states that people attribute more value to things that they own and more inclined to retain them than obtaining the same object when they do not possess it. Based on this concept, value is not absolute but perceptual in nature, and perceived ownership would affect perceived value. The endowment effect is supported by the loss aversion stating that losses have a stronger impact than gains. The asymmetry between the impact of positive and negative expectations or experiences on oneself is traced back to evolution. Organisms that had considered dangers as more important than opportunities had a better chance of survival and reproduction. Providing a condition in which children can keep the rewards after treatment only if they behave cooperatively may be more powerful reinforcement than the traditional conditioning. Up to the authors' knowledge, except for limited studies that applied the endowment effect in creating the health policies, it has not been used in the medical field for behavioral management.

Behavioral priming is referred to as the influence of different stimuli such as words, sounds, smells, colors, and pictures on the various cognitive constructs and memory, which in turn impact the behaviors. Overall, primes are classified into two categories based on how an individual percept them, subliminal and conscious. That being said, the influence of both types of primes is mostly outside one's awareness. Several studies in the past decades showed that people can be induced to behave in certain ways such as acting socially or unsocially, walking faster or slower, and being accurate or inaccurate as a result of priming outside of their consciousness. Moreover, some new studies even used the effect of superhero priming on social behaviors and found that exposing individuals to superhero images provokes prosocial activity. Although the influence of the behavioral priming was documented in previous studies, there are still disputes about the underlying mechanisms of the priming effect. The traditional concept supports the enhanced accessibility to memory and psychological constructs that active behaviors related to certain stereotypes. However, neglecting the situational factors and other moderators led to failure in the replication of the effect of primes in some recent studies. Therefore, the new approach toward behavioral priming states that different situational factors play roles in making decisions and behaviors as well. The new approach does not undermine the unconscious effect of the prime on behaviors but emphasizes on considering the situational factors as well as the individuals' characteristics in interpreting the effects.

Besides the inductive effect of environmental forces and primes on behaviors, personality traits can be reliable predictors of decisions and behaviors as well. Personality traits are considered as a reference point and a moderator for different behaviors. This is true, especially in uncertain situations, the presence of weak environmental forces, or extremity of a person in a particular trait. Moreover, personality traits can have an impact on how individuals infer and suffer from pain and consequently, the related behaviors. Some studies reported a meaningful relationship between personality and pain perception. The five-factor theory of personality (FFT): Neuroticism (N), Extraversion (E), Openness (O), Agreeableness (A) and Conscientiousness (C) is a model which takes into account the relationship between personality and health. Furthermore, a recent systematic review found that despite the common belief, the personality traits are not permanent and can be changed through experiences. Therefore, assessing personality traits may not only have predictive value but may be employed to help with the treatment procedure.

Hypothesis:

Up to the authors' knowledge, no study has implemented the concept of endowment effect for behavioral management in the medical or dental field. Besides that, the behavioral priming has not been used in the dental field as well. The hypothesis is that implementing these two concepts can help to improve pediatric patients' cooperation during dental injections.

Objectives:

1. To investigate the priming effect of superhero posters as stimuli on the behaviors of pediatric patients during the dental injection
2. To compare the two scenarios of giving rewards to pediatric patients, i.e., before starting the treatment (endowment effect) and after finishing the treatment (positive reinforcement), in order to investigate their impact on children behaviors during the dental injection
3. To investigate the moderating role of personality traits on the behaviors of pediatric patients during dental injection
4. To investigate the moderating effect of age, gender, and family income on the behaviors of pediatric patients during dental injection

Proposed Methodology and Research Plan:

The children in mixed dentition period will participate in this clinical trial. The participants will be selected consecutively of patients refereeing to a specific dental clinic. Before beginning the dental procedures or any interventions, all the parents' of children will be asked to provide a consent form and if they agree and complete the form, then they will be asked to fill out the short form of the hierarchical personality inventory for children (HiPIC-30). The randomized block randomization method will be used to ensure the equal sample size in each group based on the interventions. Half of the children will be seeing images of the superheroes on the dental unit screen for five minutes while waiting for the dental procedure to start. If the patient is a boy, images of three popular male superheroes such as Superman, Batman, and Spiderman will be shown. If the patient is a girl, images of Wonder-woman, Batgirl, and Cat-woman will be shown. The other half of the patients will see no images on the screen. Before starting the treatment procedure, children in each group will again be subdivided into two other groups. One group will be given reward before starting the procedure, but they will be told they only can keep the reward after the treatment if they have a cooperative behavior during the dental procedure (endowment effect). The reward will be put on a tray where the child can see it throughout the dental procedure. The other group will not receive any reward at the beginning, but they will be told that they will be given a reward if they cooperate during the dental procedure to evaluate the effect of positive reinforcement. Children are free to choose their reward, as it has been shown gender, age, and cultural differences may affect the children choice. However, some small toys of superheroes will be included among the awards to test whether seeing the images of superheroes affect the award choice or not. To comply with the ethics, all children will receive the reward after treatment irrespective of their behavior.

The children behavior (outcome measure) during the dental injection will be recorded and scored later using Frankl's scale for general behavior by two examiners to prevent subjectivity of measurement. The children recordings from the time of needle penetration until taking out the needle will be scored. Frankl's scale helps to categorize the behavior into four levels. To reduce the confounding effects, dentists who wear the same coat for every dental visit will perform the dental examinations and procedures. Moreover, the dental office where the examinations take place will be the same for all children.

Sample Size Calculation and Data Analysis:

The sample size will be calculated using GPower v3.1.9 software for the independent t-test. Considering a medium to large effect size=0.6, α level=0.05, statistical power (1-β)=0.85, the sample size of n=102 will be obtained. However, as the outcome measure is non-parametric, an additional 4 samples will be recruited. Therefore, 106 participants will be needed for the non-parametric test. However, considering 10% for drop-outs and missing data, the final sample size will reach 117. The main effects of interventions i.e. priming effect and reward system will be evaluated with the Mann-Whitney test. Moreover, using ordinal logistic regression, the predictive value of the main variables and moderators for children's behavior will be calculated.

Potential Outcomes and Expected Research Contribution:

Patient management in pediatric dentistry is a matter of great importance to achieve a successful and effective treatment. Injecting the children patients is one of the most challenging steps for dentists which determine the cooperation of a child for the rest of the treatment. The techniques proposed in this study are straightforward to apply in dental settings with a minimum of the cost. We hope that the results of this interdisciplinary approach be a step forward for future projects. The results will contribute to an interdisciplinary approach toward patient management and a treatment plan that let practitioners manage their time more efficiently, and also increase the chance of children's acceptable behaviors and cooperation during a dental visit and attendance in follow-up sessions.

ELIGIBILITY:
Inclusion Criteria:

1. children who need dental treatment and injection
2. children between 6 to 12 years old
3. children without severe or chronic orofacial pain
4. children without chronic systemic disease
5. children who had not dental injection in the past six months
6. children whose parents are present at the operation room

Exclusion Criteria:

1. being a non-English speaker
2. children whose parents are not willing their child to be videotaped or participate in the study
3. history of post-traumatic stress disorders or specific phobia related to the dental settings
4. children who supposed to have a dental extraction
5. children who stay in the waiting room for more than one hour

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2019-06-12 (Actual); Primary Completion 2019-06-12 (Actual); Study Completion 2019-06-12 (Actual)

PRIMARY OUTCOMES:
Behavior of the children during the dental injection | Approximately 20 seconds
  Accessing behavior of children during dental injection (from the time of needle penetration until taking out the needle) using Frankl's scale which categorize behaviors into four levels i.e. 1. definitely negative 2. negative 3. positive 4. definitely positive

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Moharrami, DDS, Principal Investigator — University of Alberta

IPD SHARING:
Plan to Share IPD: No